CLINICAL TRIAL: NCT05039086
Title: Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines (DREAM)- PDE5
Brief Title: Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines (DREAM) - PDE5
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Rutgers University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Rishi J. Desai, Assistant Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2019A010961-8
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Phosphodiesterase 5 Inhibitors; Endothelin Receptor Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PDE5 inhibitors: Exposure group
  Interventions: Drug: PDE5 inhibitor
- Endothelin receptor antagonists: Reference group
  Interventions: Drug: Endothelin Receptor Antagonists

INTERVENTIONS:
Drug: PDE5 inhibitor — PDE5 inhibitors (sildenafil, tadalafil) claim is used as the exposure group.
  Groups: PDE5 inhibitors
Drug: Endothelin Receptor Antagonists — Endothelin receptor antagonists (bosentan, ambrisentan, macitentan) claim is used as the reference group.
  Groups: Endothelin receptor antagonists

SUMMARY:
This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the DREAM Study of Brigham and Women's Hospital. DREAM is led by Dr. Madhav Thambisetty, MD, PhD, Chief of the Clinical and Translational Neuroscience Section, Laboratory of Behavioral Neuroscience, National Institute on Aging (NIA) intramural research program. This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication using healthcare claims data.

ELIGIBILITY:
Please see https://docs.google.com/spreadsheets/d/19NwmDi8xwWjzXqhSLPDTg4CKHt5UDQXuwCnZwY8jCS8/edit?usp=sharing or Appendix A for full code and algorithm definitions.

Medicare timeframe: 2008 to 2018 (end of data availability).

Inclusion Criteria:

* 1. Aged > 65 years on the index date
* 2. No prior use of PDE5 inhibitors (sildenafil, tadalafil) and endothelin receptor antagonists (bosentan, ambrisentan, macitentan) anytime prior to cohort entry date
* 3. Enrollment in Medicare Part A, B, and D with no HMO coverage for 365 days prior to and including cohort entry date

Exclusion Criteria:

* 1. Prior history of dementia measured anytime prior to cohort entry date
* 2. No prior history of pulmonary arterial hypertension recorded in the 365 days prior to cohort entry date
* 3. Prior history of nursing home admission in the 365 days prior to the cohort entry date

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: This study will employ a new user, active comparator, observational cohort study design comparing PDE5 inhibitors (sildenafil, tadalafil) to endothelin receptor antagonists (bosentan, ambrisentan, macitentan). The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of study drugs (cohort entry/index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).
Sampling Method: Non-Probability Sample
Enrollment: 13021 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Thambisetty, MD, PhD, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PDE5 Inhibitors | Endothelin Receptor Antagonists
Started (Study cohort before 1:1 propensity score matching) | 9968 | 3053
Completed (Study cohort after 1:1 propensity score matching) | 2888 | 2888
Not Completed | 7080 | 165

BASELINE CHARACTERISTICS:
Population: Study cohort after 1:1 propensity score matching
Groups:
- Total: Total of all reporting groups
Arm/Group | PDE5 Inhibitors | Endothelin Receptor Antagonists | Total
Number analyzed (Participants) | 2888 | 2888 | 5776
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 2888 | 2888 | 5776
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.87 (6.43) | 73.84 (6.15) | 73.86 (6.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1999 | 1990 | 3989
  Male | 889 | 898 | 1787
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2293 | 2311 | 4604
  Black | 421 | 411 | 832
  Asian | 51 | 53 | 104
  Hispanic | 48 | 46 | 94
  Native American | 11 | 11 | 22
  Other | 49 | 41 | 90
  Unknown | 15 | 15 | 30
Dementia risk factors [Count of Participants; unit: Participants]
  Diabetes | 1180 | 1145 | 2325
  Obesity | 911 | 918 | 1829
  Hypertension | 2587 | 2595 | 5182
  Coronary artery disease | 2136 | 2150 | 4286
  Depression | 515 | 537 | 1052
  Anxiety | 466 | 465 | 931
  Bipolar disorder | 28 | 32 | 60
  Schizophrenia | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Time to Dementia Onset
Description: Time to dementia onset includes: Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Please refer to uploaded protocol for full definition.
  Analysis 1-'as-treated' follow-up approach: In this approach, we followed patients from cohort entry until treatment discontinuation or switch to the comparator treatment, insurance disenrollment, death, or administrative endpoint (December 2018). Treatment discontinuation was defined as occurring 90 days after the expected days supply.
  of the most recently filled prescription to accommodate suboptimal adherence during treatment periods.
  Analysis 2-'as-started' follow-up approach incorporating a 6-month 'induction' period.
  Analysis 3-incorporating a 6-month 'symptoms to diagnosis' period Analysis 4-high-specificity outcome definition
  Study accessed Medicare files (Jan 2008-Dec 2018) between September 1, 2021 to October 4, 2022.
Time Frame: Median follow up times: 1) 168 days (exp), 151 days (ref) 2) 693 days (exp), 720 days (ref) 3) 382 days (exp), 358 days (ref) 4) 169 days (exp), 151 days (ref)
Population: Study cohort after 1:1 propensity score matching
Measure: Number (95% Confidence Interval); unit: Incidence rate per 1000 person year
Arm/Group | PDE5 Inhibitors | Endothelin Receptor Antagonists
Number analyzed (Participants) | 2888 | 2888
Incidence rate per 1000 person year
  Analysis 1 | 17.9 [13.5 to 23.4] | 18.8 [14.3 to 24.3]
  Analysis 2 | 19.8 [15.2 to 25.4] | 19.9 [15.3 to 25.4]
  Analysis 3 | 15.1 [10.2 to 21.4] | 22.6 [16.5 to 30.1]
  Analysis 4 | 5.2 [3 to 8.4] | 4.7 [2.7 to 7.8]

ADVERSE EVENTS:
Time Frame: 'As-treated' follow-up approach - Median follow-up days of 168 (for PDE5 inihibitors) and 151 (for endothelin receptor antagonists)
Description: Our study did not capture Serious Adverse Events.
Arm/Group | PDE5 Inhibitors | Endothelin Receptor Antagonists
All-Cause Mortality (participants affected / at risk) | 327/2888 | 407/2888
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2888 | 0/2888

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT05039086/Prot_SAP_001.pdf